CLINICAL TRIAL: NCT02633839
Title: A Phase 1 Study of the Safety and Levodopa Pharmacokinetics Following Single Dose Administration of CVT 301 (Levodopa Inhalation Powder) in Smoking and Non-Smoking Adults
Brief Title: A Study of the Safety and Levodopa Pharmacokinetics Following Single Dose Administration of CVT 301 (Levodopa Inhalation Powder) in Smoking and Non-Smoking Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVT-301-007
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Smoking
Keywords: Adults
MeSH Terms: conditions — Smoking | interventions — Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adults who smoke (Experimental): Day -1, subjects begin pre-treatment of oral dose regimen of carbidopa every 8 hours.
  Day 1, subjects receive a final dose of carbidopa and 1 hour later, a single dose of CVT-301.
  Interventions: Drug: CVT-301; Drug: Carbidopa
- Adults who don't smoke (Experimental): Day -1, subjects begin pre-treatment of oral dose regimen of carbidopa every 8 hours.
  Day 1, subjects receive a final dose of carbidopa and 1 hour later, a single dose of CVT-301.
  Interventions: Drug: CVT-301; Drug: Carbidopa

INTERVENTIONS:
Drug: CVT-301 — Levodopa inhalation powder, will be supplied in capsules containing levodopa (l-dopa), designed to deliver to the lung using the CVT-301 inhaler.
Drug: Carbidopa — Administered orally according to the carbidopa dosing schedule.
  Other Names: Lodosyn ®

SUMMARY:
This is an open label, parallel group study to evaluate the pharmacokinetics (PK) and safety of a single dose of CVT-301 in smoking and non-smoking adults.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18 to 32 kg/m2;
* Forced expiratory volume in one second (FEV1) ≥80% of predicted for race, age, sex, and height;
* FEV1/FVC (forced vital capacity) ratio ≥70%;
* Smokers are defined as those currently smoking at least 10 cigarettes/day for at least 12 months with a positive urinary cotinine result and with no past (within 5 years) or present history of intrinsic lung disease (e.g. asthma, chronic obstructive pulmonary disease [COPD], chronic bronchitis, or other relevant conditions);
* Non-smokers are defined as those who never smoked or were exposed to less than 1 pack year within at least 12 months and with a negative urinary cotinine result.

Exclusion Criteria:

* Subject who is not surgically sterile or female subject who is less than 2 years postmenopausal, and who does not agree to use a highly effective birth control method during the study and up to 3 months after the last dose of investigational product;
* Any flu-like syndrome or other respiratory infections within 2 weeks prior to the Screening Visit;
* History of chronic obstructive pulmonary disorder (COPD) requiring intermittent or continuous use of any oral or inhaled medication therapy within last 3 years;
* Renal impairment as defined by a calculated creatinine clearance of ≤ 80 mL/minute;
* History of syncope within the last 6 months.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | within 30 min prior to CVT-301 dose administration and specified time points up to 24 hours post-dose
Time to maximum observed plasma drug concentration (tmax) | within 30 min prior to CVT-301 dose administration and specified time points up to 24 hours post-dose
Area under the plasma concentration versus time curve (AUC) | within 30 min prior to CVT-301 dose administration and specified time points up to 24 hours post-dose

SECONDARY OUTCOMES:
Change in pulmonary function | within 90 min prior to CVT-301 dose and at specified time points up to 24 hours post-dose
  Pulmonary function will be measured by spirometry using the guideline specified by the Third National Health and Nutrition Examination Survey (NHANES III)
Number of subjects with Adverse Events (AEs) including Serious AEs | up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Harald Murck, MD, PhD, Study Director — Acorda Therapeutics
Locations (2):
- United States (2):
  - Site 001, Daytona Beach, Florida
  - Site 002, Dallas, Texas